CLINICAL TRIAL: NCT05611294
Title: A Visual Outcome Comparison of Topography Guided LASIK Versus Small Incision Lenticule Extraction: A Prospective Contralateral Eye Study
Brief Title: Contralateral Study of Topography Guided LASIK Versus Small Incision Lenticule Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoopes Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDRR-CON2022
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Myopia; Astigmatism
Keywords: refractive surgery; myopia; astigmatism; excimer laser; femtosecond laser; VARIO Topolyzer; Lenticule
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Contralateral Eye to Eye Comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Topography-Guided LASIK (Active Comparator): Subjects receive Topography-Guided LASIK surgery on one eye.
  Interventions: Device: Topography Guided LASIK Surgery
- Small Incision Lenticule Extraction (Active Comparator): Subjects receive Small Incision Lenticule Extraction surgery on one eye.
  Interventions: Device: Small Incision Lenticule Extraction Surgery

INTERVENTIONS:
Device: Topography Guided LASIK Surgery — LASIK surgery, using corneal topography data in treatment profile, to correct myopia or myopia with astigmatism refractive error.
  Arms: Topography-Guided LASIK
Device: Small Incision Lenticule Extraction Surgery — Corneal lenticule formation using a femtosecond laser, with subsequent lenticule extraction, to correct myopia or myopia with astigmatism refractive error.
  Arms: Small Incision Lenticule Extraction

SUMMARY:
This study evaluates differences in postoperative visual outcomes between patients receiving Topography-Guided LASIK in one eye and Small Incision Lenticule Extraction in the other eye.

DETAILED DESCRIPTION:
This is a prospective, randomized, simultaneous, contralateral eye study including at least 42 patients undergoing refractive correction surgery. Patients will be selected from the Hoopes Vision patient population after a preliminary refractive evaluation has been completed. Patients who express an interest in the study will be consented. After informed consent has been obtained and the patient has completed a screening exam and met all study criteria they will be considered enrolled. Randomization will ensure 50% of Right Eyes will receive Topography-Guided LASIK and 50% of Right Eyes will receive Small Incision Lenticule Extraction. Subjects will be given postoperative care instructions and medications following standard of care practices. Subjects will return for a 1-day, 1-week, 1-month, 3-month, and 12-month visit. Retreatments may only occur after all postoperative study visits have been completed and/or the subject has exited the study. At the preliminary screening visit, 1-month, 3-month, and 12-mont postoperative visits, patients will complete a Patient Participant Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22-50 at the time of consent
2. Diagnosis of myopia or myopia with astigmatism with Preop manifest spherical equivalent of refraction of ≥ -2.00 and ≤ -9.00 D
3. Preop Spherical component of ≥ -2.00 and ≤ -8.00 D
4. Refractive Cylinder of ≤ -3.00 D
5. BCVA of 20/20 or better in each eye
6. Subjects must have a stable refraction which is defined as change in spherical equivalent no greater than 0.50 D comparing screening visit manifest refraction to previous refractions over one year period prior to surgery. (spectacle Rx, or contact lens Rx)
7. Subjects who are contact lens wearers must have hard or gas permeable lenses discontinued for at least 4 weeks and soft lenses discontinued for at least 5 days prior to the preoperative screening evaluation. Hard or gas permeable lens wearers must not return to contact lens use before surgery and soft lens wearers must discontinue use at least 5 days before surgery.
8. Acceptable topography and baseline examination results for refractive procedures as determined by Principal Investigator or Co-Investigator
9. Surgical plan includes treatment target for emmetropia in both eyes and no monovision.
10. Subject is capable and willing to use postoperative medications as prescribed.
11. Subject has ability to successfully complete all preoperative and postoperative questionnaires, testing, and exam visits.
12. Subjects are willing and able to return for all postoperative examinations.

Exclusion Criteria:

1. Clinically significant dry eye on clinical examination as determined by the investigator
2. Irregular astigmatism, keratoconus, keratoconus suspect, or abnormal corneal topography
3. History of corneal dystrophies or guttata
4. History of herpetic keratitis or active disease
5. History of prior refractive surgery
6. History of glaucoma or glaucoma suspect
7. History of uncontrolled diabetes, unstable hypertension, or unstable autoimmune disease.
8. Females who are pregnant, breast-feeding, or intend to become pregnant any time during the course of the study as determined by verbal inquiry.
9. The Principal Investigator has determined the subject not to be a good candidate for the study

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity | 12 months
  Percentage of eyes with Uncorrected Visual Acuity of 20/20 or better
Corrected Visual Acuity | 12 months
  Percentage of eyes with Corrected Visual Acuity of 20/20 or better

SECONDARY OUTCOMES:
Predictability of Intended Outcome | 12 months
  Percentage of eyes with refractive error within +/- 0.50 D MRSE and +/- 1.00 D MRSE of intended correction

CONTACTS AND LOCATIONS:
Overall Officials: Majid Moshirfar, MD, Principal Investigator — Hoopes Vision
Locations (1):
- Hoopes Vision, Draper, Utah, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers outside of those participating in this specific study.

REFERENCES:
- [Derived] Moin KA, Manion GN, Pandiri S, Hoopes PC, Moshirfar M. Three-Month Comprehensive Outcomes of Topography-Guided LASIK Versus Keratorefractive Lenticule Extraction (KLEx): A Prospective Contralateral Study. Ophthalmol Ther. 2024 Aug;13(8):2265-2284. doi: 10.1007/s40123-024-00987-y. Epub 2024 Jul 1. PMID 38951314